CLINICAL TRIAL: NCT00302926
Title: B195: Effect of Diet-Induced Energy Deficit and Body Fat Reduction on Inflammatory Markers in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Dansk Droge A/S, Industrigrenen 10, 2635 Ishøj, Denmark (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KF01-107/02
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2006-03-15 (Estimated); Status verified 2006-03

CONDITIONS: Obesity
Keywords: Weight loss; obesity; energy restriction
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Maintenance

INTERVENTIONS:
Procedure: energy restriction and maintenance

SUMMARY:
Aim: To dissociate the effects on plasma concentrations of the inflammatory marker c-reactive protein of a negative energy balance and a reduction in body fat stores. Secondly to compare CRP with fibrinogen and interleukin-6 (IL-6).

DETAILED DESCRIPTION:
Background:

Previous epidemiological studies have associated elevated levels of acute phase proteins, mainly C-reactive protein, with cardiovascular diseases (CVD) and cardiac death. Levels of several cy-tokines and acute phase proteins as CRP, haptoglobin and fibrinogen have been found associated with elevated body fat and the risk of diseases associated to the metabolic syndrome.

Method:

Thirty-six otherwise healthy obese subjects (BMI: 34.23.2 kg/m2, age: 43.410.5 y) participated in a 20-week controlled dietary intervention divided into 4 periods. Weight reduction was induced by an 8-week low caloric diet (LCD) (3.4 MJ/d) followed by a 4-week weight stable maintenance program (M1). Subsequently, they underwent another 4-week LCD (4.2 MJ/d) followed by a final 4-week weight stable maintenance diet (M2). Blood samples and anthropometrical measures were assessed at baseline and after each of the four periods (8, 12, 16 and 20 weeks).

ELIGIBILITY:
Inclusion Criteria:

* 41 participants (20 men, 21 women) were included in the study. They were between 24-62y, healthy, non-athletic, weight stabile (< 3 kg in last 2 mo) but overweight to obese (BMI: 28-40 kg/m2).

Exclusion Criteria:

* evidence of metabolic or systemic diseases other than obesity. Frequent use of medication, a systolic blood pressure >165 mmHg and diastolic blood pressure >95 mmHg.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-09; Study Completion 2003-06

PRIMARY OUTCOMES:
Weight loss
C-reactive protein
cardiovascular diseases markers
obesity
energy restriction

CONTACTS AND LOCATIONS:
Overall Officials: Anita Belza, MSci, Principal Investigator — Department of human Nutrition, The Royal Veterinary and Agricultural University, Denmark
Locations (1):
- Anita Belza, Frederiksberg, Denmark